CLINICAL TRIAL: NCT03385083
Title: Clinical Outcomes in Chronic Low Pain Back Utilizing Activity Trackers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB approval lapsed
Sponsor: New York Institute of Technology (Other)
Responsible Party: Principal Investigator, Hallie Zwibel, Assistant Professor, New York Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BHS-1292
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain | interventions — Referral and Consultation

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACTIVITY TRACKER (Experimental): Subjects in Cohort A will receive standard of care treatments in addition to a Fitbit Flex 2 activity tracker for six weeks and recommendation for daily step counts at initial visit. Cohort A will then meet with researchers via telehealth at 2 weeks and 4 weeks with researchers to review step counts and reaffirm targets. Subjects in Cohorts A will be reassessed in person at the conclusion of the six week period.
  Interventions: Behavioral: Step count monitoring with consulting; Device: Fitbit tracker
- Control (Placebo Comparator): Subjects in Cohort B will receive standard of care treatments in addition to a Fitbit Flex 2 activity tracker for six weeks and recommendation for daily step counts at initial visit. Subjects in Cohorts B will be reassessed in person at the conclusion of the six week period.
  Interventions: Behavioral: Step count monitoring without consultation; Device: Fitbit tracker

INTERVENTIONS:
Behavioral: Step count monitoring with consulting — Subject counseled on step counts at initial visit and 2 and 4 weeks
  Arms: ACTIVITY TRACKER
Behavioral: Step count monitoring without consultation — Subject counseled on step counts at initial visit
  Arms: Control
Device: Fitbit tracker — Fitbit tracker given to participant

SUMMARY:
This is a randomized controlled study to assess the effects of activity monitors, with telehealth follow ups, on the treatment of chronic low back pain subjects.

DETAILED DESCRIPTION:
This is a randomized controlled study to assess the effects of activity monitors, with telehealth follow ups, on the treatment of chronic low back pain subjects. Subjects with low back pain will present for evaluation to the NYIT Academic Health Care Center. Once serious complications have been ruled out and a diagnosis of chronic low back pain has been made, subjects will be informed about this proposed study and asked if they would like to participate. Voluntary subjects will then be consented by designated investigators. The subjects will then be randomized into either the activity tracker and telemedicine follow up group or the control group.

Once enrolled, all subjects will complete the study as outlined in the procedures. It will involve the use of several validated assessment tools. Following the initial visit, subjects in both groups will return in 6 weeks for reassessment. Subjects in the experimental group will additionally be given an activity tracker and have 2 telemedicine visits at 2 and 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years age and younger than 75 years of age
* Subjects evaluated and found to have low back lasting longer than 3 months

Exclusion Criteria:

The subject suffers from any of the following:

* Foot drop
* Recent diagnosis of malignancy
* Recent infection
* Saddle anesthesia
* Urinary or bowel incontinence
* Progressive neuromotor or sensory loss

  * The subject is unable to complete the assessment tools
  * The subject is pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Oswestry Low Back Pain Disability Questionnaire | 6 weeks
  Back pain assessment tool

SECONDARY OUTCOMES:
Step counts | 6 weeks
  Number of steps per day

CONTACTS AND LOCATIONS:
Locations (1):
- NYIT, Old Westbury, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Shared upon request
Supporting Information: Study Protocol
Time Frame: 1 year